CLINICAL TRIAL: NCT04479813
Title: Role of Sympathetic Activation in Ischemia Reperfusion Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Perth Hospital (Other)
Responsible Party: Principal Investigator, Dr Markus Schlaich, Principal Investigator, Royal Perth Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: REG 15-021
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Central Sympathetic Nervous System Diseases
Keywords: Ischemia; re-perfusion; Remote conditioning
MeSH Terms: conditions — Ischemia | interventions — moxonidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No conditioning + placebo (Experimental): Participants will be given placebo to take orally 20 minutes prior to the first endothelial function measurement without conditioning tests.
  Interventions: Other: placebo
- No conditioning + moxonidine (Experimental): Participants will be given moxonidine to take orally 20 minutes prior to the first endothelial function measurement without conditioning tests.
  Interventions: Drug: Moxonidine 0.2 MG
- Remote pre-conditioning + placebo (Experimental): Participants will be given placebo to take orally 20 minutes prior to the first endothelial function measurement with conditioning tests.
  Interventions: Other: placebo
- Remote pre-conditioning + moxonidine (Experimental): Participants will be given moxonidine to take orally 20 minutes prior to the first endothelial function measurement with conditioning tests.
  Interventions: Drug: Moxonidine 0.2 MG

INTERVENTIONS:
Drug: Moxonidine 0.2 MG — Subjects will be allocated to undergo conditioning or non conditioning assigned in a randomized order. Participants will be given placebo or 0.2mg of Moxonidine to take orally 20 minutes prior to the first endothelial function measurement.
  Arms: No conditioning + moxonidine; Remote pre-conditioning + moxonidine
Other: placebo — Subjects will be allocated to undergo conditioning or non conditioning assigned in a randomized order. Participants will be given placebo or 0.2mg of Moxonidine to take orally 20 minutes prior to the first endothelial function measurement.
  Arms: No conditioning + placebo; Remote pre-conditioning + placebo

SUMMARY:
This study is designed to assess the effect of forearm ischemia-reperfusion injury on sympathetic nerve activity. To determine whether reduced sympathetic responsiveness is a contributor to the protective effects of remote ischemic preconditioning. In addition it will assess whether pharmacologic inhibition of the sympathetic nervous system can ameliorate ischemia reperfusion injury induced endothelial dysfunction.

DETAILED DESCRIPTION:
This is a randomized single blind study where subjects will be allocated to undergo one of the 4 protocols. Participants will be given placebo or 0.2mg of Moxonidine to take orally 20 minutes prior to the first endothelial function measurement.

This medication acts by reducing the activity of nerves believed to be involved in the conditioning process. The placebo pill, designed to have no effect, will be used as a comparison. Comprehensive tests will occur which include Microneurography, Endothelial function ,Blood Sampling, Temporary block of arm blood flow and Remote conditioning

ELIGIBILITY:
Inclusion Criteria:

* healthy males, not on any medication, free of any history of metabolic, cardiovascular or cerebrovascular disease.

Exclusion Criteria:

* smoker

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 50 healthy male volunteers (25 aged 18-30 years and 25 aged 60-75 years)
Enrollment: 46 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
change in muscle sympathetic nerve activity | 1 day
  Muscle sympathetic nerve activity assessed by microneurography

SECONDARY OUTCOMES:
Endothelial Function using the EndoPat2000 device | 2 days
  Endothelial Function testing involves the measurement of pulse amplitude from the tip of each index finger at rest and after a period of occlusion using an arm cuff that is manually inflated to a level above that of the participant's Blood Pressure (BP).

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schlaich, MD,FAHA,FESC, Principal Investigator — Royal Perth Hospital
Locations (1):
- Dobney Hypertension Centre, Perth, Australia